CLINICAL TRIAL: NCT01020812
Title: Phase II Study of Combination Stereotactic Body Radiotherapy (SBRT) With Transarterial Chemo-Embolization (TACE) for Unresectable Hepatocellular Carcinoma
Brief Title: Combination SBRT With TACE for Unresectable Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: enrollment was too low
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel T. Chang, Associate Professor of Radiation Oncology (Radiation Therapy), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP0024; SU-09112009-3882 (Other: Stanford University)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Carcinoma, Hepatocellular; Hepatobiliary Neoplasm; Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiotherapy (SBRT) (Experimental): SBRT will be delivered on Varian's linear accelerator with On-Board Imaging (OBI) capabilities. The tumor will be tracked with the ethiodol material from the TACE procedure, and respiratory gating will be used to minimize motion due to respiration. Treatment will be given in either 3 or 5 fractions . SBRT will take place after the treatment planning and within 12 weeks of the last TACE procedure.
  Doses: 45 Gy at 15 Gy/fraction , 36 Gy at 12 Gy/fraction, 45 Gy at 9 Gy/fraction, 40 Gy at 8 Gy/fraction
  Interventions: Procedure: TACE; Procedure: SBRT

INTERVENTIONS:
Procedure: TACE — Standard of Care
  Other Names: Transcatheter arterial chemoembolization; Transarterial Chemoembolization
Procedure: SBRT — Standard of Care
  Other Names: stereotactic body radiotherapy

SUMMARY:
To determine the efficacy and toxicity of TACE combined with SBRT

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third most deadly cancer in the world. It is primarily seen in areas where hepatitis is endemic, such as Asia, but other risk factors include alcoholic cirrhosis.

Outcome of this disease is poor, mostly due to the fact that >80% of patients present with unresectable disease. Surgery or transplantation remain the only curative options. For the vast majority of patients who are unresectable, a variety of treatment options are available, including transarterial chemo-embolization (TACE), radiofrequency ablation, radioactive microspheres, microwave coagulation, laser-induced thermotherapy, and percutaneous alcohol injection, all of which have similar survival rates. Stereotactic body radiotherapy (SBRT) for unresectable HCC is a relatively new treatment option made available because of great improvements in diagnostic imaging and radiation delivery techniques. Although follow-up is limited, results show encouraging local control rates. Some investigators have combined TACE with fractionated radiotherapy as a means of intensifying local therapy, with some evidence of benefit.

TACE remains the dominant mode of local therapy for unresectable HCC. However, recurrence rates are high. The recent randomized trial suggests that a combination of local therapy (TACE and radiofrequency ablation [RFA]) is superior to either therapy alone, providing proof of principle that combined local treatment is most likely more effective for HCC. Because SBRT is rapidly becoming an accepted local therapy for hepatic lesions, its role in treating HCC needs to be further defined. Studies combining TACE and external beam radiotherapy have shown encouraging results, so the logical next step is to combine TACE with SBRT, which delivers a radiobiologically more intensive dose of radiation. However, toxicity data are lacking, since this combination has not been previously reported.

We propose to conduct a trial of trans-arterial chemo-embolization (TACE) and SBRT for unresectable HCC.

ELIGIBILITY:
Inclusion -

* Liver tumors treatable by SBRT not to exceed 10cm in greatest axial dimension.

  * 800 cc of uninvolved liver
  * Patients may have additional hepatic lesions if they are <3cm and can be treated with TACE or RFA.
* Age > 18 years old
* Albumin > 2.4 g/dL.
* Total bilirubin < 3 mg/dL.
* INR ≤ 1.5.
* Creatinine < 2.0 mg/dL.
* Confirmed hepatocellular carcinoma by one of the following:

  * Histopathology
  * Two radiographic techniques (out of US, MRI, CT, Angiography) that confirm a lesion >2 cm with arterial hypervascularization
  * One radiographic technique that confirms a lesion >2 cm with arterial hypervascularization and an elevated AFP
* Hepatic lesion in patients for whom surgical resection is not possible or would not result in an opportunity for cure
* Tumor(s) <10cm
* Eastern Clinical Oncology Group performance status 0, 1 or 2
* No prior surgery, chemotherapy, or radiation for the current tumor
* Patients placed on the liver transplant registry are eligible for this trial, but will be withdrawn from the protocol if they receive liver transplantation.
* TACE done prior to study enrollment is allowed if there were no more than 3 procedures within an 18 week period and SBRT can begin within 12 weeks of the last TACE procedure.

Exclusion -

* Prior radiotherapy to the upper abdomen
* Prior TACE, RFA, or liver transplant
* Tumor(s) ≥ 10cm
* Large esophageal varices without band ligation
* Active GI bleed or within 2 weeks of study enrollment
* Ascites refractory to medical therapy
* Contraindication to receiving radiotherapy
* Women who are pregnant
* Administration of any systemic cytotoxic agents within the last 12 months
* Presence of extrahepatic metastases
* Participation in another concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT and TACE: SBRT will be delivered on Varian's linear accelerator with On-Board Imaging (OBI) capabilities. The tumor will be tracked with the ethiodol material from the TACE procedure, and respiratory gating will be used to minimize motion due to respiration. Treatment will be given in either 3 or 5 fractions . SBRT will take place after the treatment planning and within 12 weeks of the last TACE procedure.
  Doses: 45 Gy at 15 Gy/fraction , 36 Gy at 12 Gy/fraction, 45 Gy at 9 Gy/fraction, 40 Gy at 8 Gy/fraction
  TACE: Standard of Care
  SBRT: Standard of Care
Period: Overall Study
Arm/Group | SBRT and TACE
Started | 11
Completed | 8
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Stereotactic Body Radiotherapy (SBRT): SBRT will be delivered on Varian's linear accelerator with On-Board Imaging (OBI) capabilities. The tumor will be tracked with the ethiodol material from the TACE procedure, and respiratory gating will be used to minimize motion due to respiration. Treatment will be given in either 3 or 5 fractions . SBRT will take place after the treatment planning and within 12 weeks of the last TACE procedure.
  Doses: 45 Gy at 15 Gy/fraction , 36 Gy at 12 Gy/fraction, 45 Gy at 9 Gy/fraction, 40 Gy at 8 Gy/fraction
  TACE: Standard of Care
  SBRT: Standard of Care
Arm/Group | Stereotactic Body Radiotherapy (SBRT)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Local Progression of TACE and SBRT at 12 Months
Description: Freedom from local progression is defined as the time from start of treatment until the first occurrence of local progression. Local progression is defined as progression in the treated lesion according to the RECIST criteria. Progression outside the treated lesion and/or death will be considered as competing risks. The data was analyzed in a competing risk model with death as a competing risk. The outcome reported is the cumulative incidence at 12 months.
Time Frame: 12 months
Population: All patients who completed treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | SBRT and TACE
Number analyzed (Participants) | 8
proportion of participants | 0.286 [0.0310 to 0.636]
Statistical Analysis 1: Comparison: SBRT and TACE; The data was analyzed in a competitive risk model with the cumulative incidence function as the estimator. Death and other progression were competitive risks; Test type: Superiority or Other; proportion of participants = 0.286, 95% CI 2-sided [0.031 to 0.636] — The data was analyzed in a competing risk model with death as a competing risk. The proportion of 0.286 is the cumulative incidence function at 12 months

2. Secondary Outcome: To Determine the Progression-free Survival of TACE and SBRT at 18 Months
Description: Progression free survival is defined as the time from the start of treatment until the first progression or death. Progression will be defined as either local progression, disease occurring elsewhere in the liver, extrahepatic progression or clinical deterioration attributable to another underlying medical condition in the absence of clear radiographic findings of progressive disease.
Time Frame: 18 months
Population: All patients who completed the treatment
Measure: Number; unit: survival probability at 18 months
Arm/Group | SBRT and TACE
Number analyzed (Participants) | 8
survival probability at 18 months | 0.400
Statistical Analysis 1: Comparison: SBRT and TACE; The data was analyzed using the Kaplan Meier estimator; Test type: Superiority or Other; probability = 0.400 — This is the overall survival probability at 18 months

3. Secondary Outcome: To Determine the Overall Survival of TACE and SBRT at 18 Months
Description: Overall survival is defined as the time from the start of treatment until death from any cause.
Time Frame: 18 months
Population: All patients who completed treatment
Measure: Number; unit: probability
Arm/Group | SBRT and TACE
Number analyzed (Participants) | 8
probability | 0.857

4. Secondary Outcome: Median Progression Free Survival
Description: Time to progression free survival is defined as the time from randomization until either death or progression of disease. The median survival was calculated using a Kaplan Meier algorithm.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT and TACE
Number analyzed (Participants) | 8
months | 12 [3 to 20]

ADVERSE EVENTS:
Time Frame: 25 months. The adverse events for recorded for the entire study period.
Arm/Group | SBRT and TACE
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT and TACE (N=8)
Fatigue (General disorders) | 2 (2) — Grade 2 fatigue
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (2) — 2 events, 1 event of grade 3 and 1 event of grade 2 liver toxicity
transiminitis (Hepatobiliary disorders) | 1 (2) — 2 events of grade 1
colonic ulcer (Gastrointestinal disorders) | 1 (1) — Grade 2
bili increase (Hepatobiliary disorders) | 1 (2) — 2 events of grade 2

LIMITATIONS AND CAVEATS:
The low enrollment of patients led to the study being terminated before the full sample size could be reached. This resulted in a smaller than anticipated pool of patients to be analyzed and conclusions that are more difficult to generalize.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes